CLINICAL TRIAL: NCT05201118
Title: Phase I Clinical Study of a Fully Human BCMA-targeting CAR (CT103A) Combined With Selinexor in the Treatment of Patients With Relapsed/Refractory Extramedullary Multiple Myeloma
Brief Title: A Study of a Fully Human BCMA-targeting CAR (CT103A) Combined With Selinexor in Patients With Relapsed/Refractory Extramedullary Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chunrui Li (Other)
Collaborators: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chunrui Li, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR CT103A SELINEXOR001
Record Dates: First submitted 2022-01-05; First posted 2022-01-21 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Extramedullary Multiple Myeloma
Keywords: CT103A; Selinexor
MeSH Terms: interventions — selinexor; CT103A chimeric antigen receptor

STUDY DESIGN:
Intervention Model Description: The efficacy and safety, as well as the pharmacokinetic and pharmacodynamic characteristics of CT103A combined with different doses of Selinexor will be assessed in patients with relapsed/refractory extramedullary multiple myeloma. In this study, CT103A will be infused at the dose of 1.0×10^6 cells/Kg, while Selinexor was set as two dosage groups of 20 mg/week and 40 mg/week. Subjects in all dose groups received a single infusion of CT103A, and at least 1 month after the infusion of CT103A, Selinexor was administered orally once a week for one year when platelet count recovered to ≥50×10^9 /L. 8 to 10 subjects were enrolled at each dose group level, with a total of 16 to 20 subjects expected to be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT103A combined with Selinexor (Experimental): All subjects will be assigned to two Selinexor dose groups of 20 mg/week and 40 mg/week after receiving a single dose infusion of CT103A.
  Interventions: Drug: Selinexor; Drug: CT103A

INTERVENTIONS:
Drug: Selinexor — Selinexor, 20 mg/tablet, is a first-in-class, oral Selective-Inhibitor-of-Nuclear-Export (SINE) compound that impedes XPO-1which is a major nuclear export protein of macromolecular cargo frequently overexpressed in MM.
Drug: CT103A — CT103A consists of autologous T lymphocytes transduced with anti-BCMA CAR lentiviral vector that containing a unique CAR structure with a fully human single-chain variable fragment (scFv).

SUMMARY:
This study is a single-center, open Phase I study, to observe the effectiveness and safety of CT103A combined with different doses of Selinexor in patients with relapsed/refractory extramedullary multiple myeloma, and the pharmacokinetics of Selinexor and CT103A Kinetic and pharmacodynamic characteristics.

DETAILED DESCRIPTION:
In this study, two dose groups of 20 mg/week and 40 mg/week will be set for Selinexor, and the dose of CT103A is 1.0×106 cells/Kg. Subjects in all dose groups will firstly receive a single dose infusion of CT103A, at least 1 month post infusion and platelet recovery to ≥50×109/L. Then subjects began to take Selinexor once a week for one year. Each dose group level will include 8-10 subjects, and a total of 16-20 subjects are expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy all the following criteria to be enrolled in the study:

  1. age ≥18 years old, male or female.
  2. Subjects with diagnosed relapsed or refractory extramedullary multiple myeloma according to IMWG criteria and have had at least 3 prior lines of therapy
  3. Evidence of cell membrane BCMA expression, as determined by a validated immunohistochemistry (IHC) or flow cytometry of tumor tissue(e.g., bone marrow biopsies, or plasmacytoma).
  4. Subjects with extramedullary myeloma require extramedullary lesions with a maximum diameter of ≥2cm
  5. ECOG score is ≤ 2
  6. Estimated life expectancy ≥ 12 weeks.
  7. Subjects should have adequate organ function:

  <!-- -->

  1. Absolute neutrophil count (ANC) ≥1×10^9 /L; absolute lymphocyte count (ALC) ≥0.3×10^9 /L; platelets ≥50×10^9 /L; hemoglobin ≥60 g/L.
  2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×upper limit of normal (ULN); total serum bilirubin ≤ 1.5×ULN.
  3. Creatinine clearance rate (CrCl) calculated according to Cockcroft-Gault formula ≥ 40 ml/min.
  4. Fibrinogen ≥ 1.0 g/L; activated partial thromboplastin time (APTT) ≤ 1.5×ULN, prothrombin time (PT) ≤1.5×ULN.
  5. SpO2 > 91%.
  6. Left ventricular ejection fraction (LVEF) ≥ 50%. 8. The subject and his/her spouse agree to use an effective contraceptive tool or medication (excluding safety period contraception) from the date of the subject's informed consent to one year post CAR T cell infusion.

  9. Subject must sign the informed consent form approved by the ethics board in person before starting any screening procedure.

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:

  1. Subjects who are known to be resistant to Selinexor;
  2. Subjects who need to use immunosuppressive agents for a long time due to graft-versus-host disease (GVHD) or autoimmune diseases.
  3. Subjects have received any anti-cancer treatment as follows: monoclonal antibody for treating multiple myeloma within 21 days before leukapheresis, or cytotoxic therapy or proteasome inhibitors within 14 days before leukapheresis, or immunomodulatory agents within 7 days before leukapheresis, or anti-tumor treatments other than those listed above within 30 days before leukapheresis.
  4. Subjects who were receiving a used therapeutic dose of corticosteroid treatment (defined as prednisone or equivalent > 20mg) within 7 days prior to screening, except for physiological alternatives, inhalation, or topical use.
  5. Subjects with hypertension that cannot be controlled by medication
  6. Subjects with serious heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (NYHA classification ≥III), and severe arrhythmias.
  7. Subjects with systemic diseases that the investigator determined to be unstable include, but are not limited to, severe liver and kidney or metabolic diseases requiring medical treatment.
  8. Subjects with second malignancies in addition to MM within the past 5 years before the screening, exceptions to this criterion: successfully treated cervical carcinoma in situ and non-metastatic basal or squamous cell skin carcinoma, local prostate cancer after radical surgery, and ductal carcinoma in situ of the breast after radical surgery.
  9. Subjects with a history of organ transplantation.
  10. Subjects have received major surgery within 2 weeks prior to leukapheresis or plan to receive surgery during the study or within 2 weeks after the study treatment (excluding local anesthesia)
  11. Subjects participated in another interventional clinical study within 1 month before signing the informed consent (ICF).
  12. Subjects with any uncontrolled active infection needed to receive systemic therapy within 7 days before leukapheresis.
  13. Positive for any of the following tests:

      * Hepatitis B virus (HBV) surface antigen (HBsAg) or hepatitis B core antibody-positive and detectable HBV DNA in peripheral blood
      * Hepatitis C virus (HCV) antibody and hepatitis C virus RNA in peripheral blood
      * Human immunodeficiency virus (HIV) antibody
      * Cytomegalovirus (CMV) DNA
      * Treponema Pallidum antibody
  14. Pregnant or lactating women.
  15. Subjects with mental illness or consciousness disorder or disease of the central nervous system
  16. Other conditions that researchers consider inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 year post CT103A infusion
  The time from the start of CT103A treatment for the subjects to the first disease progression or death for any reason.
Objective response rate (ORR) | 1 year post CT103A infusion
  The percentage of subjects who achieved sCR、CR、VGPR、PR.
Duration of response (DOR) after administration | 1 year post CT103A infusion
  DOR will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year post CT103A infusion
  OS is measured from the date of the initial infusion of CT103A to the date of the participant's death.
Minimal Residual Disease (MRD) efficacy evaluation | 1 year post CT103A infusion
  MRD evaluation according to IMWG, including the proportion of subjects who achieved MRD negative and the duration of MRD negative.
Type and incidence of adverse events (AEs) and serious adverse events (SAEs) by dose group | 1 year post CT103A infusion
  Calculate type and incidence of adverse events (AE), serious adverse event (SAE), including those happened after lymphodepletion and after infusion, those related to study drug and lymphodepletion, or those that led to withdrawal from the study. They will also be aggregated by systematic organ classification (SOC), preferred term (PT), and severity
Pharmacokinetics - Cmax of CT103A | 1 year post CT103A infusion
  The maximum transgene level at Cmax fo CT103A
Pharmacokinetics - Tmax of CT103A | 1 year post CT103A infusion
  The maximum transgene level at Tmax fo CT103A
Pharmacokinetics - AUC0-28days of CT103A | 1 year post CT103A infusion
  Area under the curve of CT103A cells from time zero to Day 28 of CT103A
Pharmacokinetics - AUC0-90days of CT103A | 1 year post CT103A infusion
  Area under the curve of CT103A cells from time zero to Day 90 of CT103A
Pharmacokinetics of Selinexor | 1 year post CT103A infusion
  The changes of concentration of Selinexor in peripheral blood will be assessed.
PD endpoints | 1 year post CT103A infusion
  The concentration levels of CAR-T-related serum cytokines such as Ferritin and IL-6
Health-related quality of life assessment | 1 year post CT103A infusion
  HRQoL will be assessed by the European Organization for Cancer Research and Treatment Quality of Life Questionnaire (EORTC-QLQ-C30)
Appraisal of life quality | 1 year post CAR-T cell infusion
  Appraisal of life quality of the subjects will be assessed by the Quality of Life Multiple Myeloma Module Questionnaire (QLQ-MY20)
Evaluation of lymphocyte subsets | 1 year post CAR-T cell infusion
  Lymphocyte subsets will be assessed by FACS
Concentration of immunoglobulins | 1 year post CAR-T cell infusion
  The levels of Immunoglobulins in peripheral blood will be assessed to monitor changes at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Chunrui Li, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keam SJ. Equecabtagene Autoleucel: First Approval. Mol Diagn Ther. 2023 Nov;27(6):781-787. doi: 10.1007/s40291-023-00673-y. Epub 2023 Sep 2. PMID 37658205